CLINICAL TRIAL: NCT02719392
Title: A Pilot Study Investigating the Efficacy of Minocycline and N-Acetyl Cysteine for Bipolar Depression
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to limited study staff and the COVID-19 pandemic, enrollment has been paused as staff hours for this project have been reduced and reallocated to other projects.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Bipolar Clinic and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016P000447
Record Dates: First submitted 2016-03-16; First posted 2016-03-25 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Bipolar Disorder; Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Acetylcysteine; Minocycline

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Minocycline (Active Comparator): Patients in the minocycline group will take 1 minocycline (100mg) and 2 NAC placebo capsules in the morning and 1 minocycline (100mg) and 2 NAC placebo capsules in the evening for a total of 6 capsules per day over the course of the study.
  Interventions: Drug: Minocycline; Other: Placebo
- N-acetylcysteine (Active Comparator): Patients in the NAC group will take 2 NAC (500mg) capsules and 1 minocycline placebo capsule in the morning and 2 NAC (500mg) capsules and 1 minocycline placebo capsule in the evening for a total of 6 capsules per day over the course of the study.
  Interventions: Dietary Supplement: N-acetylcysteine; Other: Placebo
- Minocycline + N-acetylcysteine (Active Comparator): Patients in the minocycline NAC combination group will take 2 NAC (500mg) and 1 minocycline (100mg) capsule in the morning and 2 NAC (500mg) and 1 minocycline (100mg) capsule in the evening for a total of 6 capsules per day over the course of the study.
  Interventions: Dietary Supplement: N-acetylcysteine; Drug: Minocycline
- Placebo Control (Placebo Comparator): Patients in the placebo control group will take 2 NAC placebo capsules and 1 minocycline placebo capsule in the morning and 2 NAC placebo capsules and 1 minocycline placebo capsule in the evening for a total of 6 capsules per day over the course of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: N-acetylcysteine — NAC is an FDA-approved mucolytic (a type of drug used to relieve respiratory difficulties) and is also used for the treatment of acetaminophen toxicity.
  Arms: Minocycline + N-acetylcysteine; N-acetylcysteine
Drug: Minocycline — Minocycline is an FDA-approved antibiotic commonly used to treat bacterial infections.
  Arms: Minocycline; Minocycline + N-acetylcysteine
Other: Placebo — The placebo control is an inactive sugar pill that mimics the active comparators in appearance.
  Arms: Minocycline; N-acetylcysteine; Placebo Control

SUMMARY:
The purpose of the Pilot Study Investigating the Efficacy of Minocycline and n-acetylcysteine for Bipolar Depression is to test the effectiveness of minocycline, n-acetylcysteine, and combined minocycline and n-acetylcysteine pharmacotherapy in order to fill the gap in treatments for bipolar depression. The treatment of bipolar depression remains the greatest unmet need in the management of this lifelong and chronic psychiatric disorder.

DETAILED DESCRIPTION:
The investigators are doing this research study to find out if minocycline alone, N-acetyl cysteine (NAC) alone, or the combination of minocycline and NAC can help people with bipolar depression when added to lithium. The investigators also want to find out if minocycline, NAC, and the combination of minocycline and NAC are safe to take without causing too many side effects.

While the U.S. Food and Drug Administration (FDA) has approved minocycline to treat infections and acne and has approved NAC as a mucolytic, the FDA has not approved minocycline, n-acetylcysteine, or the combination of minocycline and n-acetylcysteine to treat bipolar depression.

This research study will compare minocycline, n-acetylcysteine, and the combination of n-acetylcysteine and minocycline to placebo. The placebo looks exactly like the other study drugs, but contains neither minocycline nor NAC. During this study participants may get a placebo instead of minocycline, n-acetylcysteine, or the combination of minocycline and n-acetylcysteine. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent and follow study procedures
2. Age > or = 18 years and < or = 65 years
3. Meets Diagnostic and Statistical Manual of Mental Disorders V (DSM-V) criteria for Bipolar Disorder Type I, which is the primary focus of treatment
4. Currently depressed, as defined by a Montgomery-Asberg Depression Rating Scale (MADRS) score of > or = 18 at screen and baseline (randomization)
5. Participants will remain on baseline mood stabilizer pharmacotherapy with lithium during the study. They will need to have been on lithium with stable therapeutic blood levels for at least two weeks prior to randomization and agree not to change medications during the study.
6. Women of child bearing potential must agree to use adequate contraception (e.g. oral contraceptives, intrauterine device, double barrier methods), if sexually active. Depo Provera is acceptable if it is started 3 months prior to enrollment. If hormonal contraceptives are used, participants must also agree to use a backup method of birth control. They will also need to understand the risks of lithium and other study treatments to the fetus and infant.

Exclusion Criteria:

1. Unwilling or unable to comply with study requirements
2. Patients who are a serious suicide or homicide risk, or currently in crisis such that inpatient hospitalization or other crisis management should take priority
3. DSM-V diagnosis of Bipolar Disorder not otherwise specified, cyclothymia, schizoaffective bipolar type
4. Primary anxiety disorders (e.g. Panic disorder, generalized anxiety disorder, post-traumatic stress disorder) or patients where the anxiety disorder is the primary focus of treatment
5. Any history of obsessive compulsive disorder (OCD) or OCD-spectrum disorders
6. Clinical or laboratory evidence of hypothyroidism; if maintained on thyroid medication must be euthyroid for at least 1 month before Visit 1
7. Subjects having failed two or more trials of somatic therapy (i.e. medications for bipolar depression or Food and Drug Administration-approved devices) during the current bipolar depressive episode
8. Drug/alcohol abuse or dependence active within the past 3 months, or current substance use disorder that requires detoxification
9. Pregnancy (as determined by urine pregnancy test)
10. Suspected or known clinically unstable systemic medical disorder including epilepsy, untreated endocrine disease, unstable angina, recent ulcers or significant esophagitis
11. Conditions which may be negatively affected by minocycline treatment, such as inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease)
12. History of significant treatment non-adherence or situations where the subject is unlikely to adhere to treatment, in the opinion of the investigator
13. Current use of minocycline or history of anaphylactic reaction or intolerance to minocycline or any component of the preparation
14. Current use of greater than 500mg of NAC/day, 200ug of selenium/day or 500 IU of Vitamin E/day
15. History of anaphylactic reaction or intolerance to NAC or any component of the preparation
16. A primary clinical diagnosis of a personality disorder, or comorbid diagnosis of antisocial or borderline personality disorder
17. A history of C. difficile colitis
18. A history of tetracycline allergy
19. Liver enzymes above the upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Illness severity on the Clinical Global Impression Scale-Bipolar Version (CGI-BP) | 8 weeks
  The CGI-BP is a modified version of the CGI designed specifically for use in assessing global illness severity and change in patients with bipolar disorder. We will use the overall severity subscale to determine outcome.

SECONDARY OUTCOMES:
Quality of life on the Quality of Life, Enjoyment, and Satisfaction Questionnaire (QLES-Q) | 8 weeks
  Assesses subjective quality of life (i.e. physical health, subjective feelings, leisure activities and social relationships).
Life satisfaction on the Longitudinal Interval Follow-up Evaluation - Range of Impaired Functioning Tool (LIFE-RIFT) | 8 weeks
  Assesses extent to which psychopathology has impacted current functioning in work, household chores, interpersonal relationships with partner, family, and friends, recreational activities, and life satisfaction.
Depression severity on the Montgomery-Asberg Depression Rating Scale (MADRS) | 8 weeks
  Assesses the severity of depressive symptoms
Mania severity on the Young Mania Rating Scale (YMRS) | 8 weeks
  Assesses the severity of mania and hypomania symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Nierenberg, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No